CLINICAL TRIAL: NCT01183299
Title: Influence of a High Salt Intake on Sodium Retention, Bone Metabolism and Acid-base Balance in Immobilised Test Subjects
Brief Title: Salty Life 7 Study: Effect of High Salt Intake on Several Physiological Systems in Immobilisation
Acronym: SL7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DLR German Aerospace Center (Other)
Collaborators: Charite University, Berlin, Germany (Other); University of Erlangen-Nürnberg (Other); University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DLR-2005049
Record Dates: First submitted 2010-06-17; First posted 2010-08-17 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Bone Metabolism; Electrolyte Metabolism; Acid-Base Metabolism; Energy Metabolism; Circulation System
Keywords: bone metabolism; salt intake; acid base balance; bed rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High salt intake (Active Comparator)
  Interventions: Other: Dietary salt intake
- Low salt intake (Placebo Comparator)
  Interventions: Other: Dietary salt intake

INTERVENTIONS:
Other: Dietary salt intake

SUMMARY:
The Salty Life 7 study aimed to examine the effect of a high salt (sodium chloride, NaCl) intake on different forms of sodium retention, acid-base balance and bone metabolism and other influenced physiological systems. Because of the fact that astronauts are a vulnerable group in this context, they were of special interest. Astronauts have a high salt intake, probably because of a reduced sense of taste, as well as an increased bone resorption resulting from the lowered mechanical load in space. In which forms sodium could be retained even without fluid retention (osmotically inactive)- contrary to the argumentation of physiological text books - and if the acid-base balance is connected to sodium chloride induced bone loss is examined in a stationary bed rest study with 8 healthy, young, male test subjects. The study consisting of 2 x 21 days is carried out at the German Aerospace Center (DLR). After an adaptation period of 4 days, test subjects are immobilised in 6° head-down tilt bed rest (simulation model for some physiological changes in space) for 14 days during which they received a high (7.7 mmol NaCl/kgBW/d) and a low salt (0.7 mmol NaCl/kgBW/d) intake in cross-over design. The form of sodium retention is investigated by the calculation of daily metabolic sodium-, water- and potassium balances and by changes in body weight. The measurements of bone formation (bAP, PINP, Osteocalcin) markers as well as bone resorption markers (CTX, NTX) supply insight into the influences of a high salt intake on bone metabolism. Blood gas analysis and ph values of 24-h urine are used to gather information about accompanying changes in the acid-base balance. Further physiological systems like energy metabolism and circulation system are also under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age: 20-35 years
* Weight: 65±85kg
* Height:180±10cm.
* Successfully completed medical & psychological screening

Exclusion Criteria:

* Drugs- and alcohol abuse
* Hyperlipidemia
* Obesity
* Renal diseases
* Participant of another study in the same time frame and 3 months before starting the study
* Blood donation within the last three months before starting the study
* Risk for thrombosis
* Smoking
* Diabetes
* Rheumatism
* Bone Fracture

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-04; Study Completion 2006-04

PRIMARY OUTCOMES:
To determine the effect of salt intake on bone metabolism in bed rest | after 14 days of high and low salt intake

SECONDARY OUTCOMES:
To determine the effect of salt intake on acid base metabolism in bed rest | after 14 days of high and low salt intake
To determine the effect of salt intake on electrolyte metabolism in bed rest | after 14 days of high and low salt intake
To determine the effect of salt intake on the circulation system in bed rest | after 14 days of high and low salt intake
To determine the effect of salt intake on energy metabolism in bed rest | after 14 days of high and low salt intake

CONTACTS AND LOCATIONS:
Overall Officials: Francisca May, Dr, Principal Investigator — German Aerospace Center (DLR)
Locations (1):
- German Aerospace Center, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Rucci N, Capulli M, Piperni SG, Cappariello A, Lau P, Frings-Meuthen P, Heer M, Teti A. Lipocalin 2: a new mechanoresponding gene regulating bone homeostasis. J Bone Miner Res. 2015 Feb;30(2):357-68. doi: 10.1002/jbmr.2341. PMID 25112732